CLINICAL TRIAL: NCT03712241
Title: A Phase I, Open-label, Randomized, 4-period Crossover Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of K-285 Compared With a Single Oral Dose of Indomethacin Capsule in Healthy Adult Volunteers
Brief Title: Evaluate the Safety, Tolerability, & Pharmacokinetics of K-285 Compared With Indomethacin Capsule in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K-285-101
Record Dates: First submitted 2018-10-01; First posted 2018-10-19 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): K-285 dose/application method A
  Interventions: Drug: K-285
- Treatment B (Experimental): K-285 dose/application method B
  Interventions: Drug: K-285
- Treatment C (Experimental): K-285 dose/application method C
  Interventions: Drug: K-285
- Treatment D (Active Comparator): Indomethacin capsule
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: K-285 — Topical
  Arms: Treatment A; Treatment B; Treatment C
Drug: Indomethacin — Capsule
  Arms: Treatment D

SUMMARY:
This study is to compare the PK parameters of multiple doses and applications of K-285 with a single dose of indomethacin capsule.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study specific evaluation is performed.
* Subject is a healthy adult male or female aged 18 to 45 years, inclusive.
* Subject has a BMI of 18 to 30 kg/m2, inclusive.
* Subject meets all inclusion criteria outlined in the clinical study protocol.

Exclusion Criteria:

* Subject has abnormal findings or assessments that are clinically noteworthy at Screening or Admission (Day -1).
* Subject has a supine blood pressure after resting for 5 minutes that is higher than 140 mm Hg systolic or 90 mm Hg diastolic, or lower than 90 mm Hg systolic or 50 mm Hg diastolic at Screening or Admission (Day -1).
* Subject has a supine heart rate after resting for 5 minutes that is outside the range of 40 to 100 beats per minute at Screening or Admission (Day -1).
* Subject does not meet any exclusion criteria outlined in the clinical study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-01-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Day 2 to Day 7 of Periods 1, 2, and 3 and Day 1 of Period 4
Area under the plasma versus concentration time curve (AUC) | Day 2 to Day 7 of Periods 1, 2, and 3 and Day 1 of Period 4

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Through study completion approximately 33 to 38 days

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided